CLINICAL TRIAL: NCT05478148
Title: COMPARISON OF THE CONVENTIONAL AND MODERN TECHNIQUES USED IN CLINICAL EVALUATION AND CLASSIFICATION OF THE GINGIVAL PHENOTYPE.
Brief Title: TECHNIQUES USED IN EVALUATION OF GINGIVAL PHENOTYPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, RASUL GULIYEV, Research Asistant, Ondokuz Mayıs University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PYO.DIS.1904.21.008
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Gingival Recession
Keywords: gingival phenotype; gingival thickness
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gingival phenotype (Experimental): A Periodontal probe was used to differentiate between thick and thin phenotypes and Color coded Biotype Probe was used to classified the phenotype as thin, moderate, thick and very thick phenotypes. Endodontic File and Florida probe were used to measure the gingival thickness.
  Interventions: Device: Gingival thickness

INTERVENTIONS:
Device: Gingival thickness — After the classification the phenotype, gingival thickness was measured with Endodontic File and Modified Florida Probe from the 3 different points. First point was the probing depth level, second one was 1mm apical to this level and third one from the 2mm apical to probing depth.

SUMMARY:
This study evaluates the 4 different techniques used in clinical measurement of gingival phenotype. 1) Tranclusency of UNC-15 Periodontal Probe, 2) Transgingival probing with Endodontic file (#20), 3)Transgingival Probing with Modified Florida Probe and 4) Translucency Colorvue Biotype Probe.

The aim of our study is to evaluate the reliability and applicability of the current examination methods recommended in order to improve the deficiencies of the traditional examination methods used in the evaluation of the gingival phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals,
* Periodontal healthy individuals with a whole mouth plaque score of 15% and a whole mouth bleeding score of less than 15%,
* Individuals who have not undergone periodontal treatment (subgingival curettage, gingivectomy, crown lengthening, etc.) in the last 6 months,
* Absence of dental compensations of skeletal malocclusion.

Exclusion Criteria:

* Individuals who smoke and have a history of smoking,
* Individuals who have undergone orthodontic treatment,
* Individuals using drugs that may cause gingival hyperplasia (immunosuppressive drugs, calcium channel blockers, anticonvulsant drugs, etc.)
* Individuals who are in pregnancy or lactation period,
* Presence of structural defects, crowns or large restorations in the maxillary anterior teeth to be measured,
* The presence of missing or supernumerary teeth in the maxillary anterior teeth to be measured,

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Feasibility and reliability of techniques | 1 day
  Comparison between the conventional techniques(Periodontal probe and Endodontic file) and modern techniques(Colorvue Biotype Probe and Modified Florida Probe) in terms of reliability and feasibility.

SECONDARY OUTCOMES:
The amount of gingival thickness and the width of the keratinized tissue | 1 day
  To determine the cut-off dimensions by evaluating the gingival thickness at 3 different points.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University Faculty of Dentistry, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No